CLINICAL TRIAL: NCT00999973
Title: Study on the Effect of Mitomycin C 0.02% on the Corneal Endothelial After Photorefractive Keratectomy in Moderate Myopia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: 8804
Record Dates: First submitted 2009-10-13; First posted 2009-10-22 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitomycin c 0.02% (Active Comparator)
  Interventions: Drug: Mitomycin C 0.02%
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mitomycin C 0.02%
  Arms: Mitomycin c 0.02%
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this study 126 eyes in 63 patients with moderate bilateral myopia and astigmatism between -3 and -5 (SE difference between two eyes should not be more than 0.75 and the residual corneal thickness>350 μ ) were entered in the study. One eye went randomly under PRK with mitomycin C 0.02% in 15 min and then the other eye went under the operation without MMC. UCVA,BCVA, refractory error after the operation and the number of endothelial cells before and after the surgery would be compared in 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 19 < age < 60
* Refractory error stabled for at least one year
* No corneal pathology
* -3 < bilateral myopia and astigmatism < -5 with no difference more than 0.75 between 2 eyes

Exclusion criteria:

* Keratoconus
* Ectatic corneal disease
* Glaucoma
* Corneal dystrophy
* Lens changes affecting the visual acuity
* Anterior or posterior uveitis
* Corneal scar

Ages: 19 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 2009-09

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran